CLINICAL TRIAL: NCT06230172
Title: Early Weaning of Infants Less Than 1800 Grams From Incubator To Crib
Brief Title: Early Weaning From Incubator To Crib
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1944411
Record Dates: First submitted 2023-10-04; First posted 2024-01-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hypothermia, Newborn; Body Temperature Changes; Newborn Thermal Injury
MeSH Terms: conditions — Hypothermia; Body Temperature Changes | interventions — Hot Temperature

STUDY DESIGN:
Intervention Model Description: The investigators will compare a retrospective control arm with a prospective intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Prospective group (>1600 grams) (Experimental): The prospective group is weaned from incubator to crib at a postnatal weight of >1600 grams following consent process.
  Interventions: Radiation: Weaning incubator (heat) at an lower postnatal weight

INTERVENTIONS:
Radiation: Weaning incubator (heat) at an lower postnatal weight — Infants in the intervention group are weaned in the same manner as the infants in the control arm; however, the wean begins at a lower postnatal weight.
  Our institutional guidelines for weaning infants from incubator to crib was unchanged for both groups.

SUMMARY:
The purpose of this study is to determine the safety and feasibility of weaning from the incubator at a lower post-natal weight at 1600 grams. Our hypothesis is that early weaning from the incubator to a crib/bassinet is safe and may result in a decrease in length of hospital stay while maintaining appropriate growth velocity. Specific outcomes the investigators will evaluate are the length of hospital stay and growth velocity at early weaning.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birth weight <1600 gm

Exclusion Criteria:

* Infants who have bradycardia (HR<80 bpm) that require stimulation for resolution.
* Infants who require phototherapy.
* Infants who require respiratory support >2 liter per minute flow by nasal cannula, oxygen need can vary between 21-100%.
* Infants with major congenital anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From birth date to hospital discharge, assessed up to 52 weeks
  Duration of hospital stay

SECONDARY OUTCOMES:
Growth velocity | From birth date to hospital discharge, assessed up to 52 weeks
  Weight gain following wean from incubator to crib

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zecca E, Corsello M, Priolo F, Tiberi E, Barone G, Romagnoli C. Early weaning from incubator and early discharge of preterm infants: randomized clinical trial. Pediatrics. 2010 Sep;126(3):e651-6. doi: 10.1542/peds.2009-3005. Epub 2010 Aug 9. PMID 20696729
- [Background] Shankaran S, Bell EF, Laptook AR, Saha S, Newman NS, Kazzi SNJ, Barks J, Stoll BJ, Bara R, Gabrio J, Childs K, Das A, Higgins RD, Carlo WA, Sanchez PJ, Carlton DP, Pavageau L, Malcolm WF, D'Angio CT, Ohls RK, Poindexter BB, Sokol GM, Van Meurs KP, Colaizy TT, Khmour A, Puopolo KM, Garg M, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health, and Human Development Neonatal Research Network. Weaning of Moderately Preterm Infants from the Incubator to the Crib: A Randomized Clinical Trial. J Pediatr. 2019 Jan;204:96-102.e4. doi: 10.1016/j.jpeds.2018.08.079. Epub 2018 Oct 15. PMID 30337189